CLINICAL TRIAL: NCT05651139
Title: The Effectiveness of Using Vibration Device to Ease Pain During Injections Into the Upper Extremity: a Randomized Controlled Trial
Brief Title: Vibration Device Effect on Post-Injection Pain in the Upper Extremity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hatan Mortada (Other Government)
Responsible Party: Sponsor-Investigator, Hatan Mortada, Co-investigator, King Saud Medical City
Organization: King Saud Medical City (Other Government)
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A3261446
Record Dates: First submitted 2022-11-14; First posted 2022-12-14 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2022-12

CONDITIONS: Injection Site Inflammation; Upper Extremity Problem
Keywords: Vibration simulation; Vibration Therapy; Post-Injection Pain; Upper extremity injection pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Receiving vibration stimulation post-injection (Experimental): Using a vibration device post-injection on the affected area.
  Interventions: Device: Electrical Vibration Device
- control group (No Intervention): No intervention will be conducted

INTERVENTIONS:
Device: Electrical Vibration Device — An electrical Vibration Massage device will be used to induce deep tissue vibration stimulation
  Arms: Receiving vibration stimulation post-injection

SUMMARY:
Background: Vibratory stimulation is one of several non-pharmacological techniques used to reduce pain. Local vibration therapy generates vibrations that can penetrate up to 6 centimeters into the tissue and is utilized to manage muscle tone, alleviate localized pain, and induce an increase in blood and lymphatic circulation. This therapy is most commonly used to treat chronic pathologies of the muscles, tendons, and joints. A few studies investigating the effects of local vibration therapy on skeletal muscles and joints have found it to be beneficial in improving joint mobility and decreasing pain. Previous reports have indicated that whole-body vibration can suppress chronic low back pain, knee osteoarthritis, and peripheral neuropathy. The aim of this study is to evaluate the effects of the application of vibration stimulation on upper extremity injection-induced pain and satisfaction.

Objectives: The purpose of this study is to assess the effect of vibration stimulation application on upper extremity injection pain and satisfaction.

Methods: An electrical massage kit that induces vibration will be used on adult patients who are scheduled to receive local anesthesia or corticosteroid injections in their upper extremities. Two validated scales will be used to first assess the pain after the injection and the patient's satisfaction following the use of the vibration device.

DETAILED DESCRIPTION:
Study design:

randomized controlled trial

Study duration:

12 months, beginning in November 2022 and ending in May 2023.

Study settings:

Data will be collected from patients coming to the plastic surgery department.

Study population: adult patients scheduled to receive local anesthesia or corticosteroid injections in their upper extremities.

Eligibility criteria: Adult patients with (ASA) physical status class 1 who are scheduled to receive local anesthesia or corticosteroid injections

Sample size:

60 adult patients who are attending plastic surgery clinic for upper extremity injections.

Ethical consideration:

The authors have no ethical or financial considerations to disclose.

Rationale for using the device:

Vibrational stimulation is a relevant treatment option for pain. It has shown promise in reducing pain in a number of musculoskeletal conditions where it has been used successfully. There aren't any randomized controlled trials that explore the effect vibration stimulation has on post-injection pain in the upper extremity.

Data collection method:

Data will be collected through a data sheet. The co-investigators will collect the data directly from the patients after the injections and measure the pain using a visual analogue scale for pain. A satisfaction visual scale is also provided to assess satisfaction with the vibration device. There will also be a control group that will receive the injections without using the vibration device. Randomization will be carried out using a coin flip.

Statistical analysis:

Data will be analyzed using SPSS 24.0 version statistical software. Descriptive statistics (mean, standard deviation, frequencies, and percentages) will be used to describe the quantitative and categorical variables. Bivariate statistical analysis will be carried out using appropriate (chi-square, student's t test, one-way analysis of variance, and Pearson's correlation) statistical test, based on the type of study and outcome variables. A p-value of <0.05 and 95% CI will be used to report the statistical significance and precision of results

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* American Society of Anesthesiologists (ASA) physical status class I
* Pain free
* Adult patients scheduled to receive local anesthesia or corticosteroid injections in their upper extremities

Exclusion Criteria:

* Those on analgesic medications
* Alcoholics, drug abusers
* Pregnant patients
* Menstruating women
* Patients with reported allergies
* Patients with acute infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
The effects of vibration on upper extremity injection-induced pain | Pain will be measured immediately after receiving the intervention (with in 2 minutes)
  Measuring the pain using the Visual Analog Scale (VAS) for pain, which is a validated tool.
  the scale measures pain from 0 (no pain) to 10 (pain as bad as it could possibly be)
The effects of vibration on injection satisfaction for upper extremity injections | The satisfaction will be measured immediately post-injection and intervention (with in 5 minutes)
  The satisfaction will be measured using Satisfaction visual analog scale, which is a validated tool.
  the scale measures the satisfaction from 0 (not satisfied) to 10 (very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University Medical City, Riyadh, Central Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided